CLINICAL TRIAL: NCT00736645
Title: A Randomized, Double Blind, Placebo Controlled Clinical Trial of L-SeMet Supplementation and Finasteride Treatment of Patients With Prostate Cancer Prior to Robotic Prostatectomy/Brachytherapy
Brief Title: Selenomethionine and Finasteride Before Surgery or Radiation Therapy in Treating Patients With Stage I or Stage II Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Roswell Park Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CDR0000611962; RPCI I 104607 (Other: Roswell Park Cancer Institute)
Record Dates: First submitted 2008-08-15; First posted 2008-08-18 (Estimated); Results first posted 2017-11-28 (Actual); Last update posted 2023-10-02 (Actual); Status verified 2023-09

CONDITIONS: Prostate Cancer
Keywords: adenocarcinoma of the prostate; stage I prostate cancer; stage II prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Selenomethionine; Finasteride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Arm I (Experimental): Patients receive oral selenomethionine and oral finasteride once daily for 4-5 weeks.
  Interventions: Dietary Supplement: selenomethionine; Drug: finasteride
- Arm II (Experimental): Patients receive oral placebo and oral finasteride once daily for 4-5 weeks.
  Interventions: Drug: finasteride; Other: placebo
- Arm III (Experimental): Patients receive oral selenomethionine and oral placebo once daily for 4-5 weeks.
  Interventions: Dietary Supplement: selenomethionine; Other: placebo
- Arm IV (Placebo Comparator): Patients receive two oral placebos once daily for 4-5 weeks.
  Interventions: Other: placebo

INTERVENTIONS:
Dietary Supplement: selenomethionine — Given orally
  Arms: Arm I; Arm III
Drug: finasteride — Given orally
  Arms: Arm I; Arm II
Other: placebo — Given orally
  Arms: Arm II; Arm III; Arm IV

SUMMARY:
RATIONALE: Selenomethionine may slow the growth of prostate cancer. Testosterone can cause the growth of prostate cancer cells. Finasteride may fight prostate cancer by lowering the amount of testosterone the body makes. Giving selenomethionine together with finasteride before surgery or radiation therapy may be an effective treatment for prostate cancer.

PURPOSE: This randomized phase II trial is studying how well selenomethionine and finasteride work when given before surgery or radiation therapy in treating patients with stage I or stage II prostate cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To investigate the effects of selenomethionine and/or finasteride on key androgen receptor signaling biomarkers (prostate-specific antigen, kallikrein 2, and NKX3.1) in prostate tissue samples from patients with stage I or II prostate cancer.

Secondary

* To analyze the effects of selenomethionine and/or finasteride on apoptosis induction in benign prostate tissue samples from these patients.

Tertiary

* To determine whether responsiveness to selenomethionine and/or finasteride is related to the level of Prx1 in prostate cancer cells.

OUTLINE: Patients are randomized to 1 of 4 treatment arms.

* Arm I: Patients receive oral selenomethionine and oral finasteride once daily for 4-5 weeks. Patients then undergo prostatectomy or brachytherapy.
* Arm II: Patients receive oral placebo and oral finasteride once daily for 4-5 weeks. Patients then undergo prostatectomy or brachytherapy.
* Arm III: Patients receive oral selenomethionine and oral placebo once daily for 4-5 weeks. Patients then undergo prostatectomy or brachytherapy.
* Arm IV: Patients receive two oral placebos once daily for 4-5 weeks. Patients then undergo prostatectomy or brachytherapy.

Blood samples are collected at baseline and on the day of prostatectomy or brachytherapy. Samples are analyzed for testosterone and 5-α-dihydrotestosterone levels by capillary gas chromatography-mass spectrometry; genetic polymorphisms in the type 2 5-α reductase gene by PCR and sequencing analyses; and selenium levels by atomic absorption spectrophotometry. Additional blood samples will be stored for future analysis of alpha and gamma tocopherol, lycopene, and other vitamin levels. Toenail samples are also collected to provide an indicator of long-term selenium status. Prostate tissue samples are collected during and after prostatectomy or prior to brachytherapy. Samples are analyzed for expression of biomarkers (e.g., prostate-specific antigen, kallikrein 2, and NKX 3.1) by quantitative RT-PCR and apoptosis by TUNEL assay, immunohistochemistry, and ELISA.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically proven adenocarcinoma of the prostate

  * Diagnosed by sextant or greater biopsy
  * Clinical stage < T3 (stage I or II) disease
* Prostate-specific antigen < 20.0 ng/mL
* Gleason score < 8
* Scheduled to undergo prostatectomy or brachytherapy

PATIENT CHARACTERISTICS:

* Life expectancy > 5 years
* No other prior malignancy (excluding nonmelanoma skin cancer) in the past 5 years
* Willing and able to take finasteride, selenomethionine, and/or placebo for 3-5 weeks prior to prostatectomy/brachytherapy

PRIOR CONCURRENT THERAPY:

* More than 1 year since prior finasteride, dutasteride, Sereona repens (saw palmetto), or any other 5-α reductase inhibitor
* No prior hormonal therapy or radiotherapy
* More than 30 days since prior and no concurrent participation in any other clinical trial involving a medical, surgical, nutritional, or life-style intervention (e.g., dietary modification or exercise)
* No concurrent selenium dietary supplement at doses > 200 mg/day, including multivitamin supplements

  * At least 30 days since > 200mg/day of prior selenium dietary supplement
* No other concurrent hormonal therapy, including 5-α reductase inhibitors (e.g., finasteride or dutasteride); anti-androgens (e.g., bicalutamide, flutamide, or ketoconazole); or luteinizing hormone-releasing hormone agonists (e.g., leuprolide acetate, goserelin acetate, or abarelix)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2008-08; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James L. Mohler, MD, Principal Investigator — Roswell Park Cancer Institute
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm A: Finasteride + Selenium Placebo: Patients receive oral placebo and oral finasteride once daily for 4-5 weeks.
  Finasteride: Given orally
  Placebo: Given orally
- Arm B: Finasteride + Selenium: Patients receive oral selenomethionine and oral finasteride once daily for 4-5 weeks.
  Selenomethionine: Given orally
  Finasteride: Given orally
- Arm C: Finasteride Placebo + Selenium Placebo: Patients receive two oral placebos once daily for 4-5 weeks.
  Placebo: Given orally
- Arm D: Finasteride Placebo + Selenium: Patients receive oral selenomethionine and oral placebo once daily for 4-5 weeks.
  Selenomethionine: Given orally
  Placebo: Given orally
Period: Overall Study
Arm/Group | Arm A: Finasteride + Selenium Placebo | Arm B: Finasteride + Selenium | Arm C: Finasteride Placebo + Selenium Placebo | Arm D: Finasteride Placebo + Selenium
Started | 13 | 15 | 14 | 13
Completed | 13 | 13 | 14 | 13
Not Completed | 0 | 2 | 0 | 0
Not completed — Adverse Event | 0 | 2 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All treated and eligible patients
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A: Finasteride + Selenium Placebo | Arm B: Finasteride + Selenium | Arm C: Finasteride Placebo + Selenium Placebo | Arm D: Finasteride Placebo + Selenium | Total
Number analyzed (Participants) | 13 | 15 | 14 | 13 | 55
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.9 (7.5) | 62.0 (7.7) | 61.2 (5.2) | 61.9 (6.8) | 60.8 (6.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0
  Male | 13 | 15 | 14 | 13 | 55
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 3 | 1 | 0 | 5
  White | 12 | 12 | 13 | 13 | 50
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Effects of Selenium and Finasteride and Their Combination on PSA Level
Description: Compare PSA levels with Finasteride Placebo + Selenium Placebo group (Arm C). The Wilcoxon Rank Sum Test was used to test the difference of PSA levels of Arm A, Arm B, Arm D with Arm C.
Time Frame: 1 year
Population: All treated and eligible patients
Measure: Median (Full Range); unit: ng/mL
Arm/Group | Arm A: Finasteride + Selenium Placebo | Arm B: Finasteride + Selenium | Arm C: Finasteride Placebo + Selenium Placebo | Arm D: Finasteride Placebo + Selenium
Number analyzed (Participants) | 13 | 15 | 14 | 13
ng/mL | 1.9 [0.8 to 2.6] | 1.9 [1.7 to 2.2] | 2.0 [1.4 to 2.7] | 2.1 [1.3 to 2.7]
Statistical Analysis 1: Comparison: Arm A: Finasteride + Selenium Placebo vs Arm C: Finasteride Placebo + Selenium Placebo; Test type: Other; p = 0.5137, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Arm B: Finasteride + Selenium vs Arm C: Finasteride Placebo + Selenium Placebo; Test type: Other; p = 0.8994, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Arm C: Finasteride Placebo + Selenium Placebo vs Arm D: Finasteride Placebo + Selenium; Test type: Other; p = 0.3463, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Effects of Selenium and Finasteride and Their Combination on Apoptosis Induction
Description: Compare cleaved caspase 3 values with Finasteride Placebo + Selenium Placebo group (Arm C). The Wilcoxon Rank Sum Test was used to test the difference of cleaved caspase 3 values of Arm A, Arm B, Arm D with Arm C.
Time Frame: 1 year
Population: All treated and eligible patients
Measure: Median (Full Range); unit: percentage of apoptotic cells
Arm/Group | Arm A: Finasteride + Selenium Placebo | Arm B: Finasteride + Selenium | Arm C: Finasteride Placebo + Selenium Placebo | Arm D: Finasteride Placebo + Selenium
Number analyzed (Participants) | 13 | 15 | 14 | 13
percentage of apoptotic cells | 0.1 [0 to 11.1] | 0 [0 to 0.7] | 0 [0 to 0.4] | 0 [0 to 0.7]
Statistical Analysis 1: Comparison: Arm A: Finasteride + Selenium Placebo vs Arm C: Finasteride Placebo + Selenium Placebo; Test type: Other; p = 0.2609, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Arm B: Finasteride + Selenium vs Arm C: Finasteride Placebo + Selenium Placebo; Test type: Other; p = 0.7504, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Arm C: Finasteride Placebo + Selenium Placebo vs Arm D: Finasteride Placebo + Selenium; Test type: Other; p = 0.9727, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Arm/Group | Arm A: Finasteride + Selenium Placebo | Arm B: Finasteride + Selenium | Arm C: Finasteride Placebo + Selenium Placebo | Arm D: Finasteride Placebo + Selenium
Serious Adverse Events (participants affected / at risk) | 0/13 | 2/15 | 1/14 | 2/13
Other Adverse Events (participants affected / at risk) | 2/13 | 3/15 | 4/14 | 3/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A: Finasteride + Selenium Placebo (N=13) | Arm B: Finasteride + Selenium (N=15) | Arm C: Finasteride Placebo + Selenium Placebo (N=14) | Arm D: Finasteride Placebo + Selenium (N=13)
Cardiac valve disease (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Postoperative ileus (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urine analysis abnormal (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A: Finasteride + Selenium Placebo (N=13) | Arm B: Finasteride + Selenium (N=15) | Arm C: Finasteride Placebo + Selenium Placebo (N=14) | Arm D: Finasteride Placebo + Selenium (N=13)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Orchitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Dysuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes